CLINICAL TRIAL: NCT05871125
Title: Identifying Ideal Reimbursement "Dose" to Reduce Clinical Trial-related Financial Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Breast Cancer Research Foundation of Alabama (Unknown); Community Foundation of Greater Birmingham Women's Breast Health Fund (Unknown)
Responsible Party: Principal Investigator, Courtney Williams, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-300009554; P30CA013148 (NIH); 0 (Other Grant/Funding Number: Community Foundation of Greater Birmingham Women's Breast Health Fund)
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving reimbursement (Experimental): Monthly reimbursement to offset trial-related expenses
  Interventions: Behavioral: Reimbursement

INTERVENTIONS:
Behavioral: Reimbursement — Patients will be dosed in cohorts of 5, with a maximum available sample size of 30. The first cohort of 5 patients will be enrolled at the first reimbursement dose level of $1000 per month for 4 months ($4000 per patient in total). At the end of the 4-month period, reimbursement dose suitability will be determined as suitable by a cumulative negative financial toxicity screen and reimbursement dose deemed acceptable and appropriate in at least 4 patients. If the reimbursement dose is found suitable, we will de-escalate the reimbursement dose for the next cohort of 5 patients. If the reimbursement dose is found unsuitable, the next cohort of 5 patients will be enrolled at the same reimbursement amount ($1000 per month for 4 months).

SUMMARY:
The goal of this clinical trial is to identify the recommended financial reimbursement amount for women with breast cancer enrolled in a clinical trial. The main questions it aims to answer are:

1. What is the recommended financial reimbursement amount in trial-enrolled women with breast cancer experiencing financial toxicity?
2. What do patients think about receiving a reimbursement for trial-incurred expenses?

Participants will receive a monthly reimbursement to compensate for their trial-incurred expenses in cohorts, which will de-escalate for the next participant cohort if patients find the reimbursement dose suitable (negative financial toxicity screen, reimbursement dose deemed acceptable/appropriate). Researchers will also use qualitative interviews to explore patient perceptions of the trial reimbursements.

DETAILED DESCRIPTION:
Our overall objective is to innovatively use a dose-finding approach to identify the recommended reimbursement amount for women with breast cancer enrolled in a clinical trial. We hypothesize that optimal reimbursement for trial-related expenses will decrease patient financial toxicity and increase trial retention. The rationale is that understanding the impact of reimbursement for trial-related costs will aid in addressing socioeconomic barriers to trial participation, thus allowing for more diversity in trial enrollment and ensuring equitable efficacy of cancer treatments when used in real-world clinical settings.

Aim 1. Identify the recommended reimbursement amount in trial-enrolled women with breast cancer experiencing financial toxicity. We propose a pilot reimbursement dose de-escalation trial (continual reassessment method design; N=30) testing a monthly reimbursement for trial-enrolled patients who screen positive for financial toxicity. We will oversample patients who are Black (50%) or residing in rural locations (50%). Monthly patient-reported financial toxicity and reimbursement acceptability and appropriateness will be captured. Reimbursement dose will start at $1000 and de-escalate if patients find the reimbursement dose suitable (negative financial toxicity screen, reimbursement dose deemed acceptable/appropriate).

Aim 2. Explore patient perceptions of trial reimbursement amounts. Using semi-structured interviews, we will explore the effects of reimbursement on specific covered and uncovered trial-related costs, financial toxicity, and current retention and future participation in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be women with breast cancer currently enrolled in the Investigation of Serial studies to Predict Your Therapeutic Response with Imaging and Molecular AnaLysis (I-SPY TRIAL 2) at the UAB Medical Oncology Clinic.

Exclusion Criteria:

* Non-English speakers
* Males
* Females without cancer
* Female cancer patients not enrolled in the I-SPY TRIAL 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who receive all reimbursements and who complete follow-up surveys (overall feasibility of intervention) | 2 years
  80% retention of patients and retained patients completing at least 75% of surveys while enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Williams, DrPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No